CLINICAL TRIAL: NCT05246904
Title: Validating a Self-fitting Hearing Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00015143
Record Dates: First submitted 2022-01-31; First posted 2022-02-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hearing and Vision Loss
Keywords: hearing aids, self-fitting
MeSH Terms: conditions — Deaf-Blind Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to arm 1 (audiologist fit) or arm 2 (self fit) first. After 2-3 weeks they will be tested and then assigned to the opposite arm.
Who Masked: Participant
Masking Description: Participants will be randomly assigned and will not know which fit is first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- audiologist arm (Active Comparator): A research audiologist will fit the participant with the hearing devices according to usual clinical best practice procedures.
  Interventions: Other: Fitting algorithm
- self-fit arm (Active Comparator): Participants will follow manufacturer's printed instructions to complete the self-hearing test using the hearing aids and a provided app to program their hearing aids.
  Interventions: Other: Fitting algorithm

INTERVENTIONS:
Other: Fitting algorithm — The best fitting algorithm will be selected by the audiologist (arm 1) or software.

SUMMARY:
Eargo, Inc. has developed a hearing aid that contains self-fitting gain software that allows adults with mild-to-moderate hearing loss to test their hearing sensitivity and program hearing aids to match their measured hearing loss. Traditionally, hearing aids are custom programmed by a hearing health professional based on a professional hearing test. This technology has the potential to improve affordability and accessibility of hearing aids for adults with mild-to-moderate hearing loss. We propose to validate Eargo's self-fitting software in a clinical trial comparing self-fitting hearing aid outcomes to the same hearing aid fit by a professional following usual clinical best practice for fitting hearing aids.

DETAILED DESCRIPTION:
The study will recruit 30-50 adults age 18 and over with mild-to-moderate hearing loss in both ears. We will aim to recruit a sample with roughly equal number of males and females and new and experienced hearing aid users (defined by any hearing aid use within the previous 6 months). Hearing loss will be measured using the results of a standard clinical hearing test.

We will use a within-subject, crossover design in which all participants will complete both field trial hearing aid conditions (self-fit and clinically fit hearing aids). The order of the field trials will be randomized across participants to account for any potential order effects. After each field trial, participants will visit the lab to complete study outcome measures, including hearing aid benefit, subjective sound quality, and speech in noise intelligibility testing.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate hearing loss ability to follow written directions,

Exclusion Criteria:

* inability to use software during first visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Abbreviated profile of hearing aid benefit | 2-3 weeks
  Survey of subjective benefit
Speech in noise test, AZ Bio sentences | Immediately after fitting
  Sentence recognition test in background noise

SECONDARY OUTCOMES:
Subjective sound quality rating | 2-3 weeks
  Participants rate the quality of sound through hearing aids

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided